CLINICAL TRIAL: NCT06712017
Title: A Descriptive, Retrospective, Single-Arm Cohort Study on the Use of Selective Internal Radiation Therapy (SIRT) with Yttrium-90 Microspheres for Unresectable Primary Hepatocellular Carcinoma (HCC) in the Chinese Population
Brief Title: Observational Study for SIR-Spheres Therapy for the Treatment of HCC Patients in China
Status: Enrolling by invitation | Type: Observational
Sponsor: GrandPharma (China) Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ST-GPN00561-CP001
Record Dates: First submitted 2024-11-14; First posted 2024-12-02 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Hepatocellular Carcinoma (HCC); Hepatocellular Carcinoma Non-Resectable
Keywords: yttrium 90; y-90; HCC; SIRT
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- adult HCC patients treated with yttrium90
  Interventions: Device: Yttrium-90 (Y-90) resin microspheres

INTERVENTIONS:
Device: Yttrium-90 (Y-90) resin microspheres — selective internal radiation therapy

SUMMARY:
Yttrium-90 (y90) Microsphere Injection Solution was approved by the NMPA in 2022. Currently, there is a lack of summary of real-world data in China. Therefore, this retrospective real-world study is intented to explore the characteristics and efficacy of HCC patients treated with y90 in China, aiming to provide reference for guiding and optimizing clinical practices and subsequent confirmatory clinical studies for the treatment of HCC patients in China.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years old;
2. confirmed diagnosis of HCC
3. treated with yttrium-90 during 2023.1.1 - 2024.6.30 and assessed at least once for tumor response within 6 months following treatment

Exclusion Criteria:

no formal exclusion criteria in a real-world study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult HCC patients treated with yttrium-90 during 2023.1.1 - 2024.6.30 and assessed at least once for tumor response within 6 months following treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
best hepatic ORR measured by mRECIST criteria | 6 months following y90 therapy

SECONDARY OUTCOMES:
ORR measured by mRECIST criteria | 6 months following y90 therapy
OS | From date of first Y90 therapy until the date of death from any cause, assessed up to 24 months
TTP | From date of first Y90 therapy until the date of first documented progression, assessed up to 24 months
  time to progression
PFS | From date of first Y90 therapy until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 6 months following y90 therapy

CONTACTS AND LOCATIONS:
Overall Officials: Xiaobin Feng, MD, Principal Investigator — Beijing Tsinghua Changgeng Hospital; Kangshun Zhu, MD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University; Yefa Yang, MD, Principal Investigator — Eastern Hepatobiliary Surgery Hospital
Locations (6):
- China (6):
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Jinan, Guangdong
  - Xi'An International Medical Center Hospital, Xi’an, Guangxi
  - No.1 Affiliated Hospital of Xian Jiaotong University, Xi’an, Shanxi
  - Beijing Tsinghua Changgung Hospital, Beijing
  - The Third Affiliated Hospital of Naval Medical University, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided